CLINICAL TRIAL: NCT03598491
Title: Feasibility of a Water-soluble Contrast Application Into Dysphagia Evaluation
Status: Completed | Type: Observational
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Hwang, Associated Professor, PhD and MD, Ulsan University Hospital
Other Study IDs: chhwang10
Record Dates: First submitted 2018-07-13; First posted 2018-07-26 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Dysphagia; Swallowing Disorder
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Iohexol: Iohexol was applied in video-fluoroscopic-swallowing study
- Barium: Barium was applied in video-fluoroscopic-swallowing study

SUMMARY:
In traditional video-fluoroscopic-swallowing study, a lipid-soluble contrast (barium sulfate) has been used more than 30 years. However, it can cause chemical pneumonitis and subsequently impair reliability of video-fluoroscopic-swallowing study if aspirated. The authors reviewed the safety and usefulness of an water soluble agent-based swallowing test.

DETAILED DESCRIPTION:
Parallel-group, case-controlled trial was conducted from September 2015 to November 2017. All the patients who referred for video-fluoroscopic-swallowing study were screened.

Based on the pre-emptive evaluation, high-risky patients were allocated to iohexol (Omnipaque)-used video-fluoroscopic-swallowing study and others were allocated to barium sulfate-used video-fluoroscopic-swallowing study.

Statistical Package for the Social Sciences 24 was used to perform statistical analysis for the data. Quantitative data were presented as mean ± standard errors.

ELIGIBILITY:
Inclusion Criteria:

* All the patients who referred for video-fluoroscopic-swallowing study

Exclusion Criteria:

* none

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the inpatients and outpatients who referred for video-fluoroscopic-swallowing study
Sampling Method: Non-Probability Sample
Enrollment: 755 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Laryngeal protection | within 1 hour after video-fluoroscopic-swallowing study
  Penetration aspiration scale (zero to eight)

SECONDARY OUTCOMES:
Oral feeding | within 1 week before video-fluoroscopic-swallowing study
  Success of Oral feeding after video-fluoroscopic-swallowing study or not

OTHER OUTCOMES:
Tracheostomy | within 1 day before video-fluoroscopic-swallowing study
  Presence of tracheostomy or not
Allergic reaction | within 2 days before video-fluoroscopic-swallowing study
  Contrast allergic reaction to the Iohexl
Symptoms of chemical pneumonitis | within 1 week before video-fluoroscopic-swallowing study
  Radiological alteration on a chest xray
Hospital stay | within 1 day after discharge
  Total days from admission to discharge
Days to discharge | within 1 day after discharge
  Total Days from video-fluoroscopic-swallowing study to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Hwang, M.D., Ph.D., Study Director — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hwang CH. Swallowing study using water-soluble contrast agents may increase aspiration sensitivity and antedate oral feeding without respiratory and drug complications: A STROBE-compliant prospective, observational, case-control trial. Medicine (Baltimore). 2022 Jul 8;101(27):e29422. doi: 10.1097/MD.0000000000029422. PMID 35801762